CLINICAL TRIAL: NCT03160001
Title: Adjuvant Use of Niclosamide With Etanercept in Rheumatoid Arthritis: Experimental and Clinical Study
Brief Title: Niclosamide With Etanercept in Rheumatoid Arthritis
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Faiq Gorial (Other)
Responsible Party: Sponsor-Investigator, Faiq Gorial, consultant, University of Baghdad
Organization: University of Baghdad (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: PRO17050001
Record Dates: First submitted 2017-05-11; First posted 2017-05-19 (Actual); Last update posted 2018-12-12 (Actual); Status verified 2018-12

CONDITIONS: Rheumatoid Arthritis (RA)
Keywords: Niclosamide; Rheumatoid arthritis; diseases activity; Efficacy; Safety
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Lactose; Niclosamide; Etanercept

STUDY DESIGN:
Intervention Model Description: 1 patient group and 1 placebo group
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Placebo and etanercept (Placebo Comparator): Placebo lactose 500mg cap twice daily with etanercept 50mg weekly for 8 weeks
  Interventions: Drug: Placebo; Drug: Etanercept
- Niclosamide and etanercept (Experimental): Niclosamide cap 500 mg twice daily with Etanercept 50mg weekly for 8 weeks
  Interventions: Drug: Niclosamide; Drug: Etanercept

INTERVENTIONS:
Drug: Placebo — Patients with active RA and receive Etanercept for 8 weeks.: Placebo lactose 500mg cap twice daily
  Other Names: Lactose
  Arms: Placebo and etanercept
Drug: Niclosamide — Patients with active RA and receive etanercept with niclosamide cap 500mg twice daily orally as adjuvant therapy for 8 weeks
  Arms: Niclosamide and etanercept
Drug: Etanercept — Etanercept 50mg weekly
  Other Names: Enbrel

SUMMARY:
Assessment of the adjuvant use Niclosamide With Etanercept in Rheumatoid Arthritis

DETAILED DESCRIPTION:
In this randomized double blind placebo-controlled pilot study (Phase I study) we will assess the efficacy and safety of adjuvant use Niclosamide With Etanercept in Rheumatoid Arthritis.

ELIGIBILITY:
Inclusion Criteria:

* Patients with RA, as defined by the American College of Rheumatology (ACR) 1987 revised criteria or ACR/EULAR 2010,
* Severly Active RA by calculating either DAS28 or SDAI or CDAI.
* Patient selected are those who started etanercept for less than 3months and still active.

Exclusion Criteria:

* Patients on nonsteroidal anti-inflammatory drugs (NSAID) 2 days before entry into this study. or methotrexate (MTX)..
* Patients with hypersensitivity or severe adverse effects to niclosamide .
* Renal impairment.
* Hepatic impairment.
* Pregnancy or a desire to become pregnant.
* Breast feeding.
* Patients with Juvenile RA [16 years old or younger].
* Patients using other conventional disease modifying antirheumatic drugs (DMARDs).
* Patients on steroid.
* Patients with coexistence other connective tissue diseases or hypothyroid disease.
* Patient with mild or inactive RA.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2017-08-15 (Actual); Primary Completion 2018-08-15 (Actual); Study Completion 2018-12-10 (Actual)

PRIMARY OUTCOMES:
Change in disease activity scale | Day 1
  Mean change of disease activity index from baseline using clinical disease activity index (CDAI).

SECONDARY OUTCOMES:
Change in disease activity score | Day 2
  Mean change of disease activity index from baseline using simplified disease activity index (SDAI).
disease activity change scale | Day 3
  Mean change of disease activity index from baseline using disease activity score 28 joints-erythrocyte sedimentation rate (DAS28-ESR).
The Change in disease activity scale | 24 hours to 48 hours day
  Mean change of disease activity index from baseline using health assessment quality of life (HAQDI).
safety of niclosamide | Day 1
  Number of participants with treatment-related adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed S Mahmood, MSc, Principal Investigator — Baghdad Teaching Hospital
Locations (1):
- Baghdad teaching Hospital, Baghdad, Iraq

IPD SHARING:
Plan to Share IPD: No